CLINICAL TRIAL: NCT01528319
Title: Open Clinical Trial of Arthroscopic Bankart Repair Using MG-1 for Dislocation of the Shoulder
Brief Title: Open-Label Study for Shoulder Dislocation Using MG-1
Acronym: MG-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-1
Record Dates: First submitted 2012-01-15; First posted 2012-02-08 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Shoulder Dislocation
Keywords: Arthroscopic Bankart repair; Suture anchor; Shoulder dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MG-1 (Experimental): Arthroscopic Bankart repair is applied for glenohumeral instability using MG-1
  Interventions: Device: MG-1

INTERVENTIONS:
Device: MG-1 — Being embedded in the area of glenohumeral instability by arthroscopic Bankart repair method.

SUMMARY:
To evaluate the efficacy and safety of arthroscopic Bankart repair using MG-1 for dislocation of shoulder

ELIGIBILITY:
Inclusion Criteria:

* Patients with dislocation of the shoulder and indicated for arthroscopic Bankart repair
* Patients of 16 years or older
* Patients who understand the contents of the study and from whom a written consent can be obtained
* Patients who can visit the hospital for follow-ups after surgery

Exclusion Criteria:

* Patients with serious complications
* Patients with comminuted fracture which may prevent fixation of the anchors
* Patients with the following diseases or conditions which may delay healing

  1. Lack of blood, infection, etc.
  2. Psychiatric disorder, alcohol poisoning, drug toxicity, etc.
  3. Tissues around the surgical site are not healthy under steroid therapy or chemotherapy
* Patients with epilepsy or bone disease (cystic change, osteopenia, etc.)
* Patients with dementia
* Patients with a history of allergy to glycolic acid, poly-L-lactic acid, β-tricalcium phosphate, polyethylene or polydioxane
* Patients who cannot undergo general anesthesia
* Patients who cannot undergo plain X-ray examination or MRI examination
* Patients with previous bone grafting in the shoulder joint
* Patients who participated in another clinical trial within past 3 months
* Patients who are pregnant or lactating. Patients who plan to be pregnant within a year
* Patients judged to be inappropriate for the study by the (sub)investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Sugaya, MD, Ph.D, Principal Investigator — Funabashi Orthopaedic Hospital
Locations (2):
- Japan (2):
  - Funabashi-shi, Chiba
  - Kobe, Hyōgo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MG-1
Started | 24
12 Weeks After Surgery | 24
Completed | 23
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | MG-1
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Region of Enrollment [Number; unit: participants]
  Japan | 24

OUTCOME MEASURES:

1. Primary Outcome: Surgery Success
Description: The rate of successful cases when surgery success is defined as "Procedure success is confirmed, the anchors are confirmed to be in the burr holes by the MRI examination, the glenohumeral ligament labral complex is maintained at the anterior edge of the glenoid cavity at 12 weeks after surgery, and there is no need of retreatment"
Time Frame: 12 weeks after surgery
Measure: Number; unit: participants
Arm/Group | MG-1
Number analyzed (Participants) | 24
participants | 23

2. Primary Outcome: Clinical Function Evaluation
Description: To evaluate the Japan Shoulder Society Shoulder Instability Score (JSS-SIS) and Rowe Score at 12 weeks after surgery
  JSS-SIS Score (subscales are summed, higher values represent a better outcome):
  * Pain (0 to 20)
  * Function (0 to 20)
  * Range of Motion (0 to 20)
  * Evaluation of X-ray findings (0 to 10)
  * Stability (0 to 30)
  Rowe Score (subscales are summed, higher values represent a better outcome):
  * Stability (0 to 50)
  * Motion (0 to 20)
  * Function (0 to 30)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MG-1
Number analyzed (Participants) | 24
units on a scale
  The JSS-SIS score | 73.7 (10.3)
  The Rowe score | 80.4 (10.7)

3. Secondary Outcome: Procedure Success
Description: The rate of successful cases when procedure success was defined as "The anchors can be inserted into the burr holes without breakage and the glenohumeral ligament labral complex can be sutured without tear of the sutures"
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | MG-1
Number analyzed (Participants) | 24
participants | 23

4. Secondary Outcome: Clinical Function Evaluation
Description: To evaluate the JSS-SIS score and Rowe score at 24 weeks after surgery
  JSS-SIS Score (subscales are summed, higher values represent a better outcome):
  * Pain (0 to 20)
  * Function (0 to 20)
  * Range of Motion (0 to 20)
  * Evaluation of X-ray findings (0 to 10)
  * Stability (0 to 30)
  Rowe Score (subscales are summed, higher values represent a better outcome):
  * Stability (0 to 50)
  * Motion (0 to 20)
  * Function (0 to 30)
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MG-1
Number analyzed (Participants) | 23
units on a scale
  The JSS-SIS score | 82.7 (7.9)
  The Rowe score | 88.9 (6.7)

5. Secondary Outcome: Number of Participants With Abnormal Changes in One or More Laboratory Tests
Description: To evaluate changes over time in each laboratory test item from before surgery to 12 and 24 weeks after surgery regarding the presence or absence of abnormal changes, causal relationship with this product and causes for development
Time Frame: 12 weeks and 24 weeks after surgery
Measure: Number; unit: participants
Arm/Group | MG-1
Number analyzed (Participants) | 24
participants | 1

6. Secondary Outcome: Adverse Event Evaluation
Description: To evaluate all undesirable events which occurred between the time of obtainment of consent and 24 weeks after surgery
Time Frame: Between the time of obtainment of consent and 24 weeks after surgery
Measure: Number; unit: participants
Arm/Group | MG-1
Number analyzed (Participants) | 24
participants | 18

ADVERSE EVENTS:
Arm/Group | MG-1
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MG-1 (N=24)
Pyogenic arthritis involving shoulder region (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MG-1 (N=24)
Cold (Infections and infestations) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No